CLINICAL TRIAL: NCT06058221
Title: Fiberoptic Intubation With Simultaneous Video-laryngoscopy Versus Through a Supraglottic Airway in Children With a Difficult Airway: a Randomized Controlled Trial
Brief Title: Hybrid Intubation Technique for Difficult Airway Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2308-024-1457
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Failed or Difficult Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid technique (Experimental)
  Interventions: Device: simultaneous videolaryngoscopy
- Supraglottic airway (Active Comparator)
  Interventions: Device: supraglottic airway

INTERVENTIONS:
Device: simultaneous videolaryngoscopy — Two specialists perform tracheal intubation, one using a video laryngoscope to expose the vocal cords and the other using a fiberoptic bronchoscope.
  Arms: Hybrid technique
Device: supraglottic airway — After inserting the supraglottic airway, the specialist performs intubation using a fiberoptic bronchoscope through the supraglottic airway.
  Arms: Supraglottic airway

SUMMARY:
To compare two hybrid techniques, flexible bronchoscopy-guided intubation with a video laryngoscope and flexible bronchoscopy-guided intubation with a laryngeal mask, that have recently shown promise as a way to increase first-attempt success rates and reduce complications in children with anticipated difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 month of age to less than 12 years of age who are expected to have a difficult intubation when undergoing routine surgery under general anesthesia.

Exclusion Criteria:

* When there is limited mouth opening, making it difficult to insert supraglottic airway ② The patient or their parents do not agree to participate in the study. ③ Other cases deemed unsuitable by the researcher

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
first attempt intubation success rate | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  The success rate of a healthcare provider's first attempt to insert a tube into a patient's airway. Intubation is defined as successful if the tube is inserted and capnography is first seen. If the fiberoptic bronchoscope comes out of the mouth, it is a failure.

SECONDARY OUTCOMES:
total intubation time (seconds) | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  Time from when the performer ends mask ventilation to when capnography first appears.
Number of intubation attempts | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  Total number of attempts to intubate, regardless of the method used (failures include bronchoscopy out of the mouth, videolaryngoscope or supraglottic airway out of the mouth, or retrying manual ventilation, even if the method is the same).
successful tracheal intubation with the allocated method | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  Whether successful in intubation according to the allocated method or not
successful tracheal intubation (Yes or No) | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  To define and confirm that "successful intubation" occurs when the endotracheal tube is successfully placed inside the trachea, capnography is visible, and surgery can proceed as a result of successful endotracheal intubation.
Nadir oxygen saturation during intubation (SpO2 value, %) | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  the minimum oxygen saturation reported during intubation periods
Oxygen reserve index during intubation (ORi™, Rainbow Signal Extraction Technology) | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  the trends of oxygen reserve index during intubation period per 5 seconds
intubation-related complication | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  Complications associated with intubation (airway injury, esophageal intubation, laryngospasm, bronchospasm, intraoral bleeding, arrhythmia, cardiac arrest).
The degree of vocal cord exposure assessed with a flexible bronchoscope. (Modified Cormack-Lehane grade, I/II/III/IV) | from induction of anesthesia to 1 minutes after intubation, about 10 minutes.
  Degree of vocal cord exposure, as determined by the Modified Cormack-Lehane grade, when a flexible bronchoscope is inserted by the anesthesiologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea